CLINICAL TRIAL: NCT06700122
Title: Clinical Comparative Evaluation of the Use of Photodynamic Therapy in Conjunction With the Use of Vitamin D in Management Stage II Grade B Periodontitis Patients: A Randomized Controlled Clinical Trial.
Brief Title: Clinical Comparative Evaluation of the Use of Photodynamic Therapy in Conjunction With the Use of Vitamin D in Management Stage II Grade B Periodontitis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Helal, Lecturer Periodontology and implantology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 391124
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-surgical periodontal therapy (SRP) and Photodynamic therapy (PDT) only (Active Comparator): * all patients will receive supragingival and sub-gingival plaque and calculus debridement (SRP) with an ultrasonic scaler and a manual universal curette where, conventional scaling and root planning (SRP) to the bottom of the pocket of 4 mm or more will be done to preserve any residual fibers attached and to avoid unintentional curettage and prevent any possible shrinkage.
  * Subgingival saline irrigation will be performed adjunctively to Sub-gingival curettage.
  * All teeth will be polished with a rubber cup. Photodynamic therapy will be done with a blue halogen curing light of wavelength 470 nm with intensity 620 mW/cm2, a continuous mode for 5 min.
  * The photosensitizer will be applied to the bottom of the periodontal pocket with the help of an applicator. After 5 min, the photosensitizer will be rinsed with saline and will be exposed to on blue halogen curing light "0" day, which will be repeated on 7th and 21st day.
  Interventions: Dietary Supplement: non-surgical periodontal therapy (SRP) and Photodynamic therapy (PDT) with systemic vitamin D
- non-surgical periodontal therapy (SRP) and Photodynamic therapy (PDT) with systemic vitamin D (Experimental): * all patients will receive supragingival and sub-gingival plaque and calculus debridement (SRP) with an ultrasonic scaler and a manual universal curette where, conventional scaling and root planning (SRP) to the bottom of the pocket of 4 mm or more will be done
  * Subgingival saline irrigation will be performed adjunctively to Sub-gingival curettage.
  * All teeth will be polished with a rubber cup. Photodynamic therapy will be done with a blue halogen curing light of wavelength 470 nm with intensity 620 mW/cm2, a continuous mode for 5 min.
  * The photosensitizer will be applied to the bottom of the periodontal pocket with the help of an applicator. After 5 min, the photosensitizer will be rinsed with saline and will be exposed to on blue halogen curing light "0" day, which will be repeated on 7th and 21st day. Serum vitamin D levels will be assessed by blood sample at baseline and 6 weeks after intervention in test group.
  Interventions: Dietary Supplement: non-surgical periodontal therapy (SRP) and Photodynamic therapy (PDT) with systemic vitamin D

INTERVENTIONS:
Dietary Supplement: non-surgical periodontal therapy (SRP) and Photodynamic therapy (PDT) with systemic vitamin D — non-surgical periodontal therapy (SRP) and Photodynamic therapy (PDT) with systemic vitamin D

SUMMARY:
Clinical Comparative Evaluation of the use of Photodynamic Therapy in conjunction with the use of Vitamin D in management Stage II Grade B Periodontitis Patients: A Randomized controlled clinical trial.

DETAILED DESCRIPTION:
This randomized clinical trial evaluates the effect of Photodynamic therapy alone with SRP versus Photodynamic therapy with SRP and Vitamin D regarding Clinical evaluation

1. Clinical attachment loss (CAL)
2. Probing pocket depth (PPD)
3. Bleeding on probing (BOP)

ELIGIBILITY:
Inclusion Criteria:

* Systemic healthy patients
* Patients aged > 25 years
* Patients suffering from stage II periodontitis with grade B were included in this study, according to 2017 world workshop classification of periodontal disease.
* Patients with interdental clinical attachment loss (CAL) of 3-4 mm with radiographic evidence of bone loss extending to coronal third of the root.
* Radiographic bone loss (RBL) will be diagnosed using periapical parallel technique using 6 radiographic images for full mouth (3- radiographic images for maxillary arch and 3- radiographic images for mandibular arch) including anterior, canine region and posterior teeth at baseline for diagnosis.
* No history of previous periodontal therapy.
* No taken medications known to interfere healing or periodontal tissue health such as anticonvulsants, calcium channel blockers, or immunosuppressant drugs.
* No previous periodontal surgery at involved sites.
* Good oral hygiene and good compliance with the plaque control instructions following initial therapy.
* Neither taken antibiotics within the last three months nor nonsteroidal anti-inflammatory drugs within the last three months
* Absence of diseases or conditions that would interfere with wound healing such as diabetes mellitus or coagulation disorders

Exclusion Criteria:

Patients taking Vitamin D as a nutritional supplement were excluded from the study

* Smoking habits
* Pregnant and lactating mothers
* Patients who have been received periodontal surgery in the study area during the last 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) | Day 0 - Week 6
  CAL will be measured form cemento- enamel junction (CEJ) to the depth of the pocket using UNC periodontal probe.
  • It will be recorded at 6 sites per tooth, the recorded readings will be used to generate mean values at each time point.

SECONDARY OUTCOMES:
Probing Pocket Depth (PPD) | Day 0 - Week 6
  PPD will be measured form free gingival margin (FGM) to the depth of the pocket using UNC periodontal probe.
Bleeding on probing (BOP) | Day 0- Week 6
  Assessment after 30 seconds after gentle brushing of the sulcus with a periodontal probe, measurement quadrant

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Helal, Principal Investigator — Cairo University
Locations (1):
- Marwa Helal, Cairo, Egypt